CLINICAL TRIAL: NCT03807284
Title: Evaluating the Feasibility of a Regaining Confidence After Stroke Course (RCAS) to Facilitate Adjustment for People With Stroke Discharged From Rehabilitation.
Brief Title: Regaining Confidence After Stroke a Feasibility Randomised Controlled Trial
Acronym: RCAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12061
Record Dates: First submitted 2019-01-10; First posted 2019-01-16 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Stroke
Keywords: Feasibility; Confidence; group intervention; Psycho-social intervention; Stroke recovery
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A parallel group two arm feasiblity randomised controlled trial with 1:1 allocation in a single centre, comparing eleven week RCAS Course in addition to usual care, to usual care alone.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor was masked to the intervention until the outcomes were complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group psycho-social course (Experimental): The intervention group received a group psycho-social course, a 2 hour, weekly, eleven week intervention delivered by a health professional working in stroke and usual care.
  Interventions: Behavioral: A group psychosocial course
- Control Group (No Intervention): Participants in the usual care control group will continue to receive all other services routinely available to them as is usual practice.

INTERVENTIONS:
Behavioral: A group psychosocial course — A 2 hour, weekly group psychosocial therapy RCAS course that aims to improve confidence and help adjustment after a stroke.
  Other Names: Regaining Confidence After Stroke Course
  Arms: A group psycho-social course

SUMMARY:
The Regaining Confidence after Stroke Course (RCAS) is a group therapy intervention to evaluate the feasibility of conducting a definitive trial, aimed to facilitate adjustment for people with stroke discharged from rehabilitation, compared with usual care. The study also aimed to evaluate the feasibility of improving mood and coping in carers of the course participants.

DETAILED DESCRIPTION:
The Regaining Confidence after Stroke Course (RCAS) is an is an eleven week group intervention that is designed to help stroke survivors when they have finished rehabilitation to improve confidence in daily life. This feasibility study aimed to evaluate the acceptability of the course in improving confidence, mood, adjustment and increasing activity levels in stroke survivors as well as improving mood and coping in their carers.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of stroke within two years
* Discharged from all other rehabilitation therapies
* Not involved in trials of other psychological interventions
* Not previously attended an RCAS course

Exclusion Criteria:

* Score of <10 on the Barthel Index (sufficiently independent to cope in a group setting)
* Score <8 on the Sheffield Screening test for Acquired Language Disorders so that participants would be able to understand the materials being presented
* Unable to speak English
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2014-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited to the trial | One year recruitment period
  Number of participants recruited to the trial
Number of participants who completed the trial | End of Study
  Number of participants who completed the trial

SECONDARY OUTCOMES:
Mood | Baseline, 3 and 6 months follow up
  GHQ-30. Mood is measured using 30 questions, each with four response scores (0=better than usual) (1= about the same) (2 =Less well than usual) (3=Much less well than usual) maximum score is 90.
Activity | Baseline, 3 and 6 months follow up
  Nottingham Extended Activity of Daily Living Scale. A ranked self-assessment of important activities after following a stroke. Scale is ranked from 0-22.
Level of Confidence | Baseline, 3 and 6 months follow up
  A Confidence after Stroke (53 item) measure. This measure uses a Likert type format with four 'Likert type' responses, from zero to three depending on a positive or negative worded item. The highest achievable score of 159 indicating a high level of confidence.
Coping | Baseline, 3 and 6 months follow up
  The COPE inventory (Coping Orientation for Problem Orientated Experiences) a 60 question measure which asks how participants deal with stress and what they do in stressful events. The inventory has 15 domains and a maximum score of 16 is achievable. A high score indicates more frequent use of the described coping strategy
Carers strain | Baseline, 3 and 6 months
  Carer Strain Index. The measure consists of 13 questions with yes or no answers. Highest score of 13 is achievable, where a high score indicates increased carer strain

REFERENCES:
- See also: Regaining Confidence after Stroke - a feasibility study. MPhil KE Hooban — http://eprints.nottingham.ac.uk/id/eprint/38848